CLINICAL TRIAL: NCT05745272
Title: Cardiovascular Risk Categories and Attaining LDL-C Targets in Middle Eastern Adults Aged 30-55 Years of Age
Acronym: CREATE
Status: Terminated | Type: Observational
Why Stopped: No enough patients to be enrolled
Sponsor: Jordan Collaborating Cardiology Group (Other)
Collaborators: The Cardiovascular Academy Group of the JCS (Unknown); The Jordan Cardiac Society (JCS) (Unknown); Istishari Hospital Department of Clinical Research (Unknown)
Responsible Party: Sponsor
Other Study IDs: CVA-G/JCS-1/2023
Record Dates: First submitted 2023-02-16; First posted 2023-02-27 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2024-01

CONDITIONS: Atherosclerotic Cardiovascular Risk; Low-density-lipoprotein (LDL) Cholesterol
Keywords: Low-density lipoprotein cholesterol (LDL-C); LDL-C targets; ASCVD risk levels; Middle East population

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Individuals evaluated for primary and secondary cardiovascular prevention have different levels of cardiovascular risk These levels of risk are the main determinants of the low-density lipoprotein cholesterol (LDL-C) target blood levels that need to be attained.

DETAILED DESCRIPTION:
Individuals evaluated for primary and secondary cardiovascular prevention fall into different levels of cardiovascular risk according to their clinical profile of having atherosclerotic cardiovascular disease (ASCVD), risk factors, and their SCORE. These levels of risk are the main determinants of the low-density lipoprotein cholesterol (LDL-C) target blood levels that need to be attained using LDL-C-lowering agents (LLA).

Contemporary studies that evaluated levels of cardiovascular risk and LDL-C goal attainment in the Middle East are scarce. A prior study (CEPHEUS LEVANT) in the Middle East demonstrated that about 1 in 4 high-risk patients reach LDL-C goals.

The current study aims at studying cardiovascular risk categories according to the 2019 ESC/EAS and 2018 ACC/AHA Guidelines, and the attainment of LDL-C treatment goals in consecutive individuals aged 18-55 years who are evaluated in tertiary care centers as inpatients or in ambulatory care settings. The above age bracket was chosen because these are the individuals most prone to acute cardiovascular events with a high prevalence of diabetes mellitus and cigarette smoking.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-55 y
* Individuals can give a history of the presence or absence of ASCVD and its risk factors

Exclusion Criteria:

* Age below 18 or older than 55
* Refusal of inability to give history on ASCVD and its risk factors

Ages: 18 Years to 55 Years | Sex: All
Age Groups: Adult
Study Population: Ambulatory care patients and in-hospital patients with any medical illness of coming for routine check ups.Age 18-55 both sexes.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2023-12-11 (Actual); Primary Completion 2023-12-15 (Actual); Study Completion 2023-12-24 (Actual)

PRIMARY OUTCOMES:
Risk level of ASCVD | 12 MONTHS
  Categorizing the patients' level of ASCVD risk by the clinical background of CVD, DM, other risk factors and 10% year risk

SECONDARY OUTCOMES:
LDL-cholesterol blood level | 12 months
  Calculating the LDL-C blood level in each patient according to the ASCVD risk category, and whether this level was attained by therapy,

CONTACTS AND LOCATIONS:
Overall Officials: Imad A. Alhaddad, MD FACC, Study Chair — Department of Cardiology, Jordan Hospital, Amman, Jordan; Ramzi Tabbalat, Study Director — Cardiology Department, Abdali Hospital; Ayman Hammoudeh, MD FACC, Principal Investigator — Department of Clinical Research, Istishari Hospital, Aman, Jordan
Locations (1):
- Istishari Hospital, Amman, Jordan

IPD SHARING:
Plan to Share IPD: Yes
CRF (CSR)
Supporting Information: CSR
Time Frame: April 2023 for 14 months